CLINICAL TRIAL: NCT00886080
Title: A Prospective Randomised Multicentre Comparison on Health Related Quality of Life: the Value of Add-on Arrhythmia Surgery in Patients With Atrial Fibrillation Undergoing Valvular and/or Coronary Bypass Surgery
Brief Title: The Effect of Arrhythmia Surgery on Quality of Life in Patients With Atrial Fibrillation Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Profileringsfonds Maastricht (Unknown)
Responsible Party: H.N.A.M. van Breugel, MD, University Hospital Maastricht
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PF 178; PF 178
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Health related Quality of Life; Add-on surgery; Ablation; Randomised controlled trial; SF-36; EuroQoL; MFI-20
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Add-on arrhythmia surgery (Experimental): Adjuvant anti-arrhythmic surgery consists of a beating heart epicardial "box" isolation of all pulmonary veins using microwave energy (Flex 4 or Flex 10 ablation probes and Microwave generator by Guidant/Afix, Fremont, CA, USA). The surgical ablation procedure is the first step during surgery and is performed before institution of cardiopulmonary bypass allowing off-pump beating heart ablation. In addition excision or exclusion of the left atrial appendage is performed in both the treated as the control group.
  Interventions: Procedure: Pulmonary vein isolation using microwave energy

INTERVENTIONS:
Procedure: Pulmonary vein isolation using microwave energy — The surgical ablation procedure is the first step during surgery and is performed before institution of cardiopulmonary bypass allowing off-pump beating heart ablation. The off-pump beating heart ablation procedure is performed according to a specific box lesion surrounding the pulmonary veins, using microwave energy. Afterwards cardiac surgery is performed as usual in both treatment arms.
  Other Names: PV-isolation

SUMMARY:
Atrial fibrillation (AF) is connected with an increased morbidity and mortality. In addition, quality of life is diminished due to palpitations, dyspnea, dizziness and syncope. AF is frequently associated with valvular and coronary disease. In the AF patients undergoing valvular or coronary surgery the arrhythmia almost always relapses. For symptom control anti-arrhythmic drugs and cardioversion are used but breakthrough arrhythmias and side effects of the drugs happen frequently. For more effective symptom control "add-on" arrhythmia surgery is being advocated. However, at present the investigators do not know whether add-on arrhythmia surgery indeed affects morbidity and quality of life.

The hypothesis being studied is that add-on arrhythmia surgery in patients with AF undergoing valvular or coronary surgery improves quality of life, establishes chronic sinus rhythm and reduces perioperative and long-term morbidity associated with AF.

DETAILED DESCRIPTION:
Multicentre prospective parallel randomised controlled trial. In total 150 patients with documented atrial fibrillation (chronic and paroxysmal), were randomly assigned by a central computer system to undergo cardiac surgery with add-on surgery or without. This assignment was blinded to patients and all medical personnel except for the surgical team during total follow up. Patients completed quality of life questionnaires, comprising the RAND 36-item Health Survey 1.0 (SF-36), Multidimensional Fatigue Inventory-20 (MFI-20) and EuroQoL (EQ-5D and VAS) at baseline and 3, 6 and 12 months following operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo valvular surgery and/ or coronary surgery,
* All patients have documented chronic atrial fibrillation of paroxysmal atrial fibrillation.
* Patients have given written informed consent.

Exclusion Criteria:

* Patients who do not speak Dutch or can not read Dutch.
* Patients with a Sick Sinus Syndrome.
* Patients with contraindications for oral anticoagulant agents.
* Incompetent to act for oneself

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2002-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Quality of life and maintenance of sinus rhythm at 1 year will be considered as primary end points. | Baseline, 3, 6, and 12 months after operation

SECONDARY OUTCOMES:
In-hospital and out-of-hospital morbidity and mortality during one year follow-up | Baseline, 1, 6 and 12 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jos G. Maessen, PhD, Study Chair — Maastricht University Medical Center
Locations (1):
- Dept. of Cardiothoracic Surgery, University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Derived] Van Breugel HN, Nieman FH, Accord RE, Van Mastrigt GA, Nijs JF, Severens JL, Vrakking R, Maessen JG. A prospective randomized multicenter comparison on health-related quality of life: the value of add-on arrhythmia surgery in patients with paroxysmal, permanent or persistent atrial fibrillation undergoing valvular and/or coronary bypass surgery. J Cardiovasc Electrophysiol. 2010 May;21(5):511-20. doi: 10.1111/j.1540-8167.2009.01655.x. Epub 2009 Nov 17. PMID 19925605